CLINICAL TRIAL: NCT04993417
Title: Comparison of Motor Imagery Technique and Mime Therapy on Facial Expressions in Facial Palsy Patients; A Randomized Clinical Trial
Brief Title: Comparison of Motor Imagery Technique and Mime Therapy on Facial Expressions in Facial Palsy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/0209 Aysha
Record Dates: First submitted 2021-07-19; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Facial Palsy
Keywords: Facial nerve palsy; Mime therapy; Motor imagery technique
MeSH Terms: conditions — Facial Paralysis; Bell Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mime Therapy along with EMS (Experimental): MT Group: Mime Therapy along with EMS
  Interventions: Other: Mime Therapy along with EMS
- Motor imagery technique along with EMS (Experimental): MIT Group: Motor imagery technique along with EMS
  Interventions: Other: Motor imagery technique along with EMS

INTERVENTIONS:
Other: Motor imagery technique along with EMS — All the subjects carried out the treatment process for a total of 3 months. During this treatment duration, the sessions were administered 3 times per week for 45 minutes, depending upon the subject's ability to focus and tiredness. The patients were mentioned to play out the emotional facial appearances for non-verbal correspondence i-e pleasure, misery, interest, appall, dread, irritation and shock. Patients were then requestedto envision himself winking, for instance, envisioning himself in a wonderful and natural social setting, at that point the patient cognitively addresses, with his eyes shut, the movement of decaying the recognized central issues, without creating any specific movement.
  Arms: Motor imagery technique along with EMS
Other: Mime Therapy along with EMS — All the subjects carried out the treatment process for a total of 3 months. During this treatment duration, the sessions were administered 3 times per week for 45 minutes, depending upon the subject's ability to focus and tiredness. Mime treatment incorporates self kneading of face and neck, breathing and relaxation works out, activities to synchronize the two sides and diminish synkinesis and for eye and lip closure per the myofascial way to deal with recovery, letter and word practices and expressive activities.
  Arms: Mime Therapy along with EMS

SUMMARY:
This project was a Randomized clinical trial conducted to compare the effects of motor imagery technique and mime therapy on facial expressions in facial palsy patients so that we can have best treatment option for patients of facial palsy. Duration was of 6 months, convenient sampling was done, subjects following eligibility criteria from Imran Idrees Teaching hospital and Idrees Hospital Sialkot, were randomly allocated in two groups via computer generated method, baseline assessment was done, MIT Group received motor imagery technique, 45 min session (3 times a week for 3 months) plus the EMS (10-15 min), while the MT Group received mime therapy 30-45 min session (3 times a week for 3 months) plus the EMS (10-15 min). Outcome measures were collected for both groups at before treatment (T0) and at the end of the treatment i-e after 3 months (T1). The outcome measures were severity of paresis, facial symmetry and intensity of depression measured by using House-Brackmann Scale, Sunnybrook Facial Grading System and Beck Depression Inventory Scale, respectively. Data was analyzed by using SPSS version 24.0.

DETAILED DESCRIPTION:
Facial palsy is due to the damage in the facial nerve that supplies the muscles of the face. Peripheral facial nerve paralysis can have various causes, such as Bell's palsy, which is the most common cause. Among secondary cause, tumors and the adverse effects of surgery for tumor pathologies such as, acoustic neuroma and facial nerve schwannoma are the most prevalent. The prognosis for FNP is complete recovery in roughly 80% of cases with Bell's palsy, whereas 15% experiences some type of permanent nerve damage, with the remaining 5% enduring severe sequelae. To this end, FNP should be treated in a multidisciplinary setting, in which physical therapy, psychological and medical or surgical interventions are integrated. The current study has compared the effects of motor imagery technique and mime therapy on facial expressions in facial palsy patients. The current study was novel in a way that there is no evidence of superiority of any rehabilitative treatment compared with another in the recovery of FNP, which was clearly determined by the current study.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral facial palsy more than 6 months
* Age 20-60 years
* House-Brackmann Scale Score ≥3
* Both genders

Exclusion Criteria:

* Pregnant women
* Psychological treatment for any psychiatric disorder
* Participants with the history of any tumor
* Diabetes

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
House-Brackmann Scale (HBS) | 12th Week
  House-Brackmann Facial Grading System comprises of six evaluations, where grade 1 addresses normal function and grade VI addresses complete loss of motion. It is quite possibly the most generally utilized scales and has been appeared to have great between rater reliability anyway its affectability to change in facial symmetry is low.

SECONDARY OUTCOMES:
Sunnybrook Facial Grading System (SFGS) | 12 Week
  SunnyBrook Facial Grading System is a 13 item evaluating scale. The framework estimates three segments of facial deviation; resting asymmetry, symmetry of voluntary activities and synkinesis. Resting lopsidedness of the eye, cheek and mouth are all things considered scored from 0 to 4 with 4 being the most uneven. Symmetry of the intentional movements; forehead wrinkle, delicate eye conclusion, open mouth grin, growl and lip pucker, are each scored from 0 to 3 with 3 being the most synkinetic, giving an all out scope of 0 to 15

OTHER OUTCOMES:
Beck Depression Inventory Scale (BDI) | 12 Week
  The 21-item Beck Depression Inventory comprises of four proclamations that depict expanding powers of depressive symptoms and incorporates substantial and intellectual emotional manifestations, everything is isolated into a scale from 0 to 3, mirroring the patient's feelings in the past fourteen days. An absolute score of each of the 21 things are created; score of 14 or above is demonstrative of depressive indications. Depressive manifestations were sorted as, minimal-moderate (14-19), moderate-severe (20-29) and severe (30-63)

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Ikram, MS, Principal Investigator — Riphah International University
Locations (1):
- Imran Idrees Teaching Hospital, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garro A, Nigrovic LE. Managing Peripheral Facial Palsy. Ann Emerg Med. 2018 May;71(5):618-624. doi: 10.1016/j.annemergmed.2017.08.039. Epub 2017 Oct 27. No abstract available. PMID 29110887
- [Background] Robinson MW, Baiungo J. Facial Rehabilitation: Evaluation and Treatment Strategies for the Patient with Facial Palsy. Otolaryngol Clin North Am. 2018 Dec;51(6):1151-1167. doi: 10.1016/j.otc.2018.07.011. Epub 2018 Sep 24. PMID 30262166
- [Background] Codari M, Pucciarelli V, Stangoni F, Zago M, Tarabbia F, Biglioli F, Sforza C. Facial thirds-based evaluation of facial asymmetry using stereophotogrammetric devices: Application to facial palsy subjects. J Craniomaxillofac Surg. 2017 Jan;45(1):76-81. doi: 10.1016/j.jcms.2016.11.003. Epub 2016 Nov 17. PMID 27939040
- [Background] Dusseldorp JR, van Veen MM, Mohan S, Hadlock TA. Outcome Tracking in Facial Palsy. Otolaryngol Clin North Am. 2018 Dec;51(6):1033-1050. doi: 10.1016/j.otc.2018.07.003. Epub 2018 Aug 29. PMID 30172554
- [Background] Greene JJ, Guarin DL, Tavares J, Fortier E, Robinson M, Dusseldorp J, Quatela O, Jowett N, Hadlock T. The spectrum of facial palsy: The MEEI facial palsy photo and video standard set. Laryngoscope. 2020 Jan;130(1):32-37. doi: 10.1002/lary.27986. Epub 2019 Apr 25. PMID 31021433
- [Background] Monsanto RD, Bittencourt AG, Bobato Neto NJ, Beilke SC, Lorenzetti FT, Salomone R. Treatment and Prognosis of Facial Palsy on Ramsay Hunt Syndrome: Results Based on a Review of the Literature. Int Arch Otorhinolaryngol. 2016 Oct;20(4):394-400. doi: 10.1055/s-0036-1584267. Epub 2016 May 30. PMID 27746846
- [Background] Joseph SS, Joseph AW, Smith JI, Niziol LM, Musch DC, Nelson CC. Evaluation of Patients with Facial Palsy and Ophthalmic Sequelae: A 23-Year Retrospective Review. Ophthalmic Epidemiol. 2017 Oct;24(5):341-345. doi: 10.1080/09286586.2017.1294186. Epub 2017 Mar 20. PMID 28319442
- [Background] Faris C, Tessler O, Heiser A, Hadlock T, Jowett N. Evaluation of Societal Health Utility of Facial Palsy and Facial Reanimation. JAMA Facial Plast Surg. 2018 Dec 1;20(6):480-487. doi: 10.1001/jamafacial.2018.0866. PMID 30178066
- [Background] D'Souza AF, Rebello SRJIJoT, Rehabilitation. Comparing the effectiveness of mime therapy and neuromuscular re-education in improving facial symmetry and function in acute Bell's palsy: a pilot randomised clinical trial. 2021;28(3):1-8.
- [Background] Park Y-K, Lee CI, Lee JH, Lee H-J, Lee Y-k, Seo J-C, et al. A Facial Chuna Manual Therapy for Peripheral Facial Nerve Palsy. 2019;36(4):197-203
- [Background] Markey JD, Loyo M. Latest advances in the management of facial synkinesis. Curr Opin Otolaryngol Head Neck Surg. 2017 Aug;25(4):265-272. doi: 10.1097/MOO.0000000000000376. PMID 28604403
- [Background] Jo YK, Lee YJ, Jeon JH, Kim YIJJoHM. Review on Clinical Studies of Facial Palsy Sequelae Treatment. 2019;28(1):1-12.